CLINICAL TRIAL: NCT06408064
Title: The Effect of Music Therapy as an Adjuvant in the Vital Signs of the Neonate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Aristizábal (Other)
Collaborators: Sanitas University (Other)
Responsible Party: Sponsor-Investigator, Claudia Aristizábal, Director, Sanitas University
Organization: Sanitas University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CEIFUS 470-24
Record Dates: First submitted 2024-04-26; First posted 2024-05-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neonatal Disease
MeSH Terms: conditions — Infant, Newborn, Diseases | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Music therapy is a non-pharmacological therapeutic intervention that will be implemented through two modalities: live and pre-recorded music. Group A will be that of patients exposed to live music, which will be carried out by a music therapist using the guitar as the only musical instrument. Instrumental lullabies will be used, which will be selected by the patients' legal guardians. Group B corresponds to patients who will be exposed to pre-recorded music, of the genre of lullabies, instrumental type, using a speaker that will be placed inside the patient's incubator. Group C will be those patients in whom no musical intervention will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Live music (Experimental): It is performed by a music therapist using the guitar as the only musical instrument. Instrumental lullabies are used, selected by the patient's legal guardian.
  Interventions: Other: Music therapy
- Pre-recorded music (Experimental): Pre-recorded music of the lullaby genre, instrumental type, using a speaker placed inside the patient's incubator.
  Interventions: Other: Music therapy
- Control (No Intervention): There will be no musical intervention.

INTERVENTIONS:
Other: Music therapy — Music therapy is a non-pharmacological therapeutic intervention that will be implemented through two modalities: live and pre-recorded instrumental lullabies music.The volume control will be conducted within the groups through the use of a decibel regulator, with a maximum volume of 70 dB. During the intervention and for a period of 30 minutes following its conclusion, singing will be prohibited by the music therapist or the parents. Both live and pre-recorded music will be instrumental in nature, lacking any lyrics.
  Arms: Live music; Pre-recorded music

SUMMARY:
The admission of a newborn to the neonatal intensive care unit (NICU) represents a potentially harmful sound environment coupled with multiple stressful events. However, a strategy such as music therapy (delivered by a trained music therapist) appears to be a non-invasive, safe, and cost-effective alternative that assists newborns in their physiological self-regulation with a beneficial effect on stabilizing neonatal vital signs, so it can be used as a complementary strategy to medical management. The aim of this study is to determine the effect of live and pre-recorded music therapy on vital sign variables in newborns older than 32 weeks hospitalized in the neonatal intensive care unit of a high-complexity health institution in Colombia.

DETAILED DESCRIPTION:
A parallel, controlled randomized clinical trial will be conducted.

Study Population: Newborns older than 32 weeks gestational age at birth hospitalized in the Neonatal Intensive Care Unit of a high-complexity health institution who meet the inclusion criteria.

Outcomes: Heart rate will be primary outcome. Respiratory rate and oxygen saturation will be secondary outcomes. The patient monitor will be utilized to measure the heart rate, respiratory rate, and oxygen saturation.

Standardization of measurements:

First, the trademarks of the medical equipment manufacturers of each of the tools that will be used (vital sign monitor and pulse oximeter) will be verified to ensure that they correspond to the same commercial brand. Since different brands may exhibit variability in standard calibration measurements within the critical range, it is important to verify that the tools are of the same brand. Secondly, it will be verified that each medical tool used has been calibrated within the previous six months, with the date of the last calibration recorded so that the device can be used during the study. Subsequently, the professional in charge of the music company will verify that the guitar to be used during the live music is in tune and suitable for use. A decibel regulator will be employed during the implementation of both pre-recorded and live music, adjusting the volume of the emitted sound. This will ensure that the decibels emitted by each research subject remain within the permitted range of 70 decibel (dB). Vital variables will be recorded at minute 0, from minute 0 to minute 10 continuously, and at 30 minutes after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with gestational age at birth greater than or equal to 32 weeks.
* Birth weight greater than or equal to 1500 grams.
* Be at least 72 hours of postnatal age.

Exclusion Criteria:

* Respiratory disturbances in the last 48 hours such as: Apnea or Brief Resolved Unexplained Events (BRUE), need for invasive mechanical ventilation
* Hemodynamic alterations in the last 48 hours such as: Hypotension (systolic, diastolic, or mean BP < P5) or hypertension (systolic, diastolic, or mean BP > P95), bradycardia (HR < 100/min), shock of any etiology, requirement for volume expanders, infusion of inotropics, vasodilators and/or prostaglandin E1.
* Neurological alterations such as: Perinatal asphyxia at birth manifested by the need for resuscitation, APGAR < 3 at 5 minutes and/or ≤ 5 at 10 minutes, and metabolic acidosis in cord gases with a potential of hydrogen (pH) < 7 and base excess (BE) < -12, hypoxic-ischemic encephalopathy, seizure syndrome for up to 48 hours after the last clinical event or alteration of the brain pattern, interventricular hemorrhage in preterm infants in the first week of diagnosis.
* Management with Extracorporeal membrane oxygenation (ECMO) and/or nitric oxide
* Temperature less than 36.5 C or greater than 37.5 C.
* Patient under pharmacological sedation or use of beta-blockers.
* Congenital heart disease, operated on or not.
* Congenital malformations
* Surgical emergencies or recovery from a surgical procedure performed within the last 48 hours.

Ages: 32 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Heart rate | The baseline measurement will be taken before the intervention, and will continue for 30 minutes during the intervention and for a further 30 minutes after the intervention has been completed.
  The measurement will be continuously quantified in terms of number of pulsations per minute continuously.

SECONDARY OUTCOMES:
Respiratory rate | The baseline measurement will be taken before the intervention, and will continue for 30 minutes during the intervention and for a further 30 minutes after the intervention has been completed.
  The measurement will be continuously quantified in terms of the number of breaths per minute.
Oxygen saturation | The baseline measurement will be taken before the intervention, and will continue for 30 minutes during the intervention and for a further 30 minutes after the intervention has been completed.
  The measurement will be continuously quantified in terms of proportion per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Johana Benavides, MSc, Study Director — Unisanitas
Locations (1):
- Clínica Universitaria Colombia, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No
When the study ends, individual participant data could be shared with the approval of the research ethics committee.

DOCUMENTS (1):
  • Study Protocol (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT06408064/Prot_000.pdf